CLINICAL TRIAL: NCT03213106
Title: Effects of Cerebellar Transcranial Magnetic Stimulation in Cerebellar Ataxias
Brief Title: Cerebellar Non-invasive Stimulation in Ataxias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Rubens Gisbert Cury, Dr Rubens Gisbert Cury, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.310.275
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Cerebellar Ataxia
Keywords: TMS; Transcranial Magnetic Stimulation; Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 5 sessions of active and sham rTMS separated by at least 4 weeks washout.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) Stimulation (Experimental): All patients will receive 5 sessions of active TMS stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham Stimulation (Sham Comparator): All patients will receive 5 sessions of active TMS stimulation
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Low frequency (1Hz) transcranial magnetic stimulation aimed to the dentate nucleus contralateral to the most symptomatic side.
  Arms: Transcranial Magnetic Stimulation (TMS) Stimulation
Device: Sham Stimulation — The stimulation coil will be placed in the same spot as the TMS stimulation, but coil will not be attached to the TMS machine.
  Arms: Sham Stimulation

SUMMARY:
Cerebellar ataxias are a group of disorders caused by cerebellar affections, for which currently no specific treatment is available. Some limited studies verified the effects of cerebellar transcranial magnetic stimulation (TMS) on ataxic symptoms, with good results. So far it is not known which patients could benefit. Our hypothesis is that cerebellar TMS could improve ataxic symptoms in some patients.

DETAILED DESCRIPTION:
Thirty patients with cerebellar ataxia will be included in our protocol. Ataxia might be due to several aetiologies, from degenerative to genetic and vascular diseases. Patients will be submitted to a neuronavigation protocol for the precise location of the dentate nucleus contralateral to the most symptomatic side. After that, participants will be randomly assigned to 5 active or 5 placebo sessions of 1Hz TMS over the located area. After the first 5 sessions and a period of at least 4 weeks washout, patients will cross over and receive other 5 sessions, active or sham. Clinical and video evaluations will be conducted before and after active and sham cluster of sessions.

ELIGIBILITY:
Inclusion Criteria:

* identification of cerebellar ataxia based on neurologic examination
* no improvement after rehabilitation
* symptoms onset of at least 6 months

Exclusion Criteria:

* Younger than 18 months
* Pregnant or breastfeeding women
* Participation in other clinical trials
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline to Post Treatment on the Scale for the Assessment and Rating of Ataxia (SARA) | Day 1 (baseline), day 5 (after 5th TMS session, active or sham), day 33 (new baseline after TMS wash out) and day 38 (after 10th TMS session, active or sham)
  Assess 8 items: gait, stance, sitting, speech, dysmetria, kinetic tremor, pro- and supinations of the hand, and the heel-shin slide. Each item is scored by the physician on a 4 to 8 numerical scale based upon the amount of dysfunction observed while performing the task. The maximum possible score for the total scale is 40. Lower scores of SARA represents better task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Rubens G Cury, MD PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franca C, de Andrade DC, Silva V, Galhardoni R, Barbosa ER, Teixeira MJ, Cury RG. Effects of cerebellar transcranial magnetic stimulation on ataxias: A randomized trial. Parkinsonism Relat Disord. 2020 Nov;80:1-6. doi: 10.1016/j.parkreldis.2020.09.001. Epub 2020 Sep 6. PMID 32920321